CLINICAL TRIAL: NCT03866369
Title: A Double-blind, Placebo-controlled, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Volunteers in Order to Define Lanifibranor (IVA337) Supra-therapeutic Dose in a Multiple Dosing Regimen
Brief Title: Multiple Ascending Dose Phase I Study in Order to Define Lanifibranor (IVA337) Supra-thjerapeutic Dose
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 337HVPK18007; 2018-003822-99 (EudraCT Number)
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy Subjects
Keywords: healthy male volunteers; multiple ascending dose; supra-therapeutic dose
MeSH Terms: interventions — Moxifloxacin; lanifibranor

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose study with 3 sequential cohorts of 12 subjects treated by Lanifibranor versus Placebo during 14 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): IMP Under investigation
  Interventions: Drug: Moxifloxacin; Drug: Placebo; Drug: Lanifibranor
- Placebo to Match (Placebo Comparator)
  Interventions: Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — Single oral dose at D-8
Drug: Placebo — Single oral dose at D-1
Drug: Lanifibranor — Single daily oral dose during 14 days
  Arms: Experimental
Drug: Placebo — Single daily oral dose during 14 days
  Arms: Placebo to Match

SUMMARY:
The study will be a double-blind, randomized, placebo-controlled, multiple ascending dose study with lanifibranor. The study will consist of up to 3 cohorts of 12 subjects each; therefore, approximately 36 subjects will be included in this study.

DETAILED DESCRIPTION:
All subject will receive first a single dose of 400 mg moxifloxacin, under open-label fasting conditions at Day -8 (assay sensitivity).

Following, all subjects also will receive a dose of placebo under open-label fasting conditions at D-1.

In the morning of Day 1, subjects will be randomized to either the investigational medicinal product (IMP) or placebo (3:1). The treatment phase last 14 days and the end of study visit will occurs within 5 to 9 days after the last dose of IMP or placebo (or at early termination)

A staggered dose approach will be applied within each subjects cohort with 48 hours of delay between subcohorts.

A sefty review committe (SRC) will review after each cohorts all available safety and PK data under blinded conditions and conclude the safety and tolerability of the dose level before proceeding to the next dose level.

ELIGIBILITY:
Main inclusion Criteria:

Subject voluntarily agrees to participate in this study and signs an IEC-approved informed consent prior to performing any of the Screening Visit procedures.

2. Males between 18 to 55 years of age (inclusive) 3. Nonsmokers (or other nicotine use) as determined by history (no nicotine use over the past 3 months) and by urine cotinine concentration (< 500 ng/mL) at the Screening Visit and admission.

4. Body mass index (BMI) between 18.0 and 29.9 kg/m2 (inclusive) at the Screening Visit.

5. Healthy with no clinically relevant deviation or finding in medical history, physical examinations, vital signs or 12-lead ECGs at the Screening Visit or admission, as applicable. Clinical laboratory values at the Screening Visit or admission should be within normal limits or judged not clinically significant as determined by the Investigator and with liver values such as:

* Alanine aminotransferase (ALT) ≤ 1.1 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 1.2 × ULN
* Gamma-glutamyltransferase (GGT) ≤ 1.5 × ULN
* Alkaline phosphatase (ALP) ≤ 1.5 × ULN

Main exclusion Criteria:

1. History or evidence of any relevant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic (e.g., diabetes), urologic, pulmonary, neurologic, psychiatric, dermatologic, renal (e.g., renal insufficiency), and/or other major disease or malignancy (e.g., bladder cancer) or present infectious disease as judged by the Investigator.
2. Subject has any surgical or medical condition that would interfere with the absorption, distribution, metabolism or excretion of drugs, or which may jeopardize the subject in case of participation in the study.

   1. Inflammatory bowel disease, peptic ulcers, gastrointestinal including rectal bleeding.
   2. Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.
   3. Pancreatic injury or pancreatitis within 12 months prior to Screening.
   4. Liver disease or liver injury as indicated by abnormally increased liver function tests. ALT, AST, GGT, ALP, and serum bilirubin will be tested at Screening.

      * Any single parameter of ALT, AST, GGT, or ALP must not exceed 1.1 x ULN and ≥ 1.2 x ULN total bilirubin.
      * Any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or serum bilirubin will exclude a subject from participation in the study.

      If necessary, laboratory testing may be repeated on one occasion (as soon as possible) prior to randomization, to rule out any laboratory error.
   5. History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or blood urea nitrogen and/or urea values, or abnormal urinary constituents (e.g. albuminuria).
   6. Evidence of urinary obstruction or difficulty in voiding
   7. History of immunodeficiency diseases.
   8. Blood levels of sodium, potassium, calcium, or magnesium outside of laboratory normal range at Screening and baseline.
   9. TSH outside of laboratory normal range at Screening.
3. Subject has any concurrent disease or condition that, in the opinion of the Principal Investigator, would make the subject unsuitable for participation in the clinical study.
4. Subject has a pulse < 50 beats per minute (bpm) or > 90 bpm; systolic BP < 90 mmHg or > 140 mmHg; diastolic BP < 50 mmHg or > 90 mmHg at the Screening Visit. One re-test is allowed, if (a) test result(s) is outside these limits.
5. Abnormal 12-lead ECG at the Screening Visit or admission, including:

   * Uncorrected QT interval ≥ 500 msec
   * QTcF > 450 msec
   * QRS interval >120 msec
   * PR interval >220 msec
   * Second or third-degree atrio-ventricular block
   * Any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant
6. Subject has clinically significant conduction disorders, significant arrhythmia or a known risk from medical history to not respond to moxifloxacin.
7. Subject has a history of additional risk factors for "Torsades de Pointe" (e.g., heart failure, hypokalemia [below the lower limit of normal], family history of Long QT Syndrome).
8. Family history of QTc prolongation or of unexplainable sudden death at < 50 years of age.
9. Any contraindication or reasons for precautionary use of moxifloxacin such as:

   * History of allergy/phototoxicity with quinolone group of drugs in the last year prior to Screening.
   * History of peripheral neuropathy.
   * History of tendinitis, tendon rupture, or clinically significant tendon injury.
   * Risk factor associated with psychiatric reactions.
   * History of seizure disorders or disease which can lower seizure threshold.
10. Subject has a history or family history of G6PD or any other congenital hemolytic anemias.
11. Subject has history of illicit drug abuse.
12. Subject has a history of drinking > 168 g pure alcohol per week (10 g pure alcohol = 259 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 2 years prior to the first admission to the clinical unit.
13. Subject has positive test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis C antibody (anti-HCV) or human immunodeficiency virus (HIV) antibodies (types 1 and 2) at the Screening Visit.
14. Subject has positive alcohol test at the Screening Visit or admission.
15. Subject has positive urine drug test (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids) at the Screening Visit or admission.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | From Baseline up to 15 days
Number of abnormal Vital signs (blood pressure, pulse) and physical exams | From Baseline up to 15 days
Number of abnormal Clinical laboratory tests (chemistry, hematology, urinalysis) | From Baseline up to 15 days
Number of abnormal 12-lead digital electrocardiograms parameters (Heart rate, QT/QTc interval, PR interval, QRS interval, RR interval) change from baseline | From Baseline up to 15 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of lanifibranor and its metabolites | 15 days
Time of maximum plasma concentration (Tmax) of lanifibranor and its metabolites | 15 days
Area under the concentration-time curve (AUC0-t) of lanifibranor and its metabolites | From Baseline up to 15 days
Number of Cardiovascular safety events | From Baseline up to 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International GmbH, Berlin, Germany